CLINICAL TRIAL: NCT01833676
Title: To Compare Effect of Sevoflurane Versus Desflurane on the Return of Protective Airway Reflexes in the Elderly Population
Brief Title: To Compare Effect of Sevoflurane Versus Desflurane on the Return of Swallowing Reflexes in the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Lee Fenky, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 901.11
Record Dates: First submitted 2013-04-06; First posted 2013-04-17 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Pulmonary Aspiration
Keywords: sevoflurane; desflurane; protective airway reflexes; elderly
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane (Active Comparator): Patient receiving Desflurane for maintenance of general anaesthesia
  Interventions: Drug: Desflurane
- Sevoflurane (Active Comparator): Patient receiving Sevoflurane for maintenance of general anaesthesia
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane
  Other Names: Sevorane
  Arms: Sevoflurane
Drug: Desflurane
  Arms: Desflurane

SUMMARY:
Anaesthesia and surgery has become more common in the elderly as the population survives longer. Anaesthesia in the elderly confers a higher risk which is related to the aging process and the diseases that accompany seniority. As such, there is a need to provide optimal anaesthetic management in order to minimize complications and risks perioperatively. One of the changes associated with ageing is the progressive decrease in protective laryngeal reflexes. Any depression of upper airway reflexes increases the chance of pulmonary aspiration and compromises the maintenance of the airway.

Desflurane is an inhalational agent strongly favored due to its lower solubility in blood, lean tissue and fat as compared to sevoflurane. This enables the agent to be quickly eliminated at the end of surgery, with minimal metabolic breakdown, thus facilitating more rapid emergence as compared to sevoflurane anesthesia in elderly undergoing general anaesthesia. McKay et al conducted a study in 2005 in US, which showed that the choice of inhalational agent itself can influence the return of protective airway reflexes. In the study, the inhalational agent sevoflurane was found to cause significant impairment of swallowing, in comparison with desflurane(1). However, the aforementioned study focussed on the general population. As such, the purpose of this study is to determine whether the choice of inhalational anesthetic (sevoflurane versus desflurane) has similar influence on the return of protective airway reflexes in the geriatric population in Malaysia, and whether the significance is greater in the elderly population.

DETAILED DESCRIPTION:
This is a prospective, double-blind, randomized controlled trial by single operator. American Society of Anaesthesiologists' classification of physical status I-II male and female patients aged 60-85 year scheduled to have general anesthesia for surgical procedures were recruited. Patients recruited will be given 20mls of water to swallow in the upright position prior to surgery after obtaining informed consent. All patients enrolled are judged to have adequate swallowing if no coughing or drooling occurred after the water passed into the mouth, and no water remained in the oropharynx upon subsequent visual inspection.

The anaesthetist in charge of the patients enrolled in the study will be given a sealed envelope containing the name of the randomised gas to be used for the patient. At the end of surgery, an observer who is blinded to the anaesthethic allocation will record the relevant data. The blinded observer determined the time to first appropriate response to command (asking the patient to 'open his/her eyes' or squeezing the observer's hand, state his/her name or state date of birth) every 30s after discontinuation of anesthetic administration and removal of LMA. Exactly 5 minutes after appropriate verbal response, patient was asked to swallow 20mls of water in a 30 degree upright position. Successful swallowing is defined as ingestion of the 20mls of water without coughing or drooling. If swallowing was successful, the study was concluded. If it was unsuccessful, the patient was asked to swallow at 5, 10, 15, 20, 25 and 30 minutes, with termination of participation after successful swallowing. A stopwatch will be used to time the duration to recovery.

A study sample size of 60 is selected, with a power of 0.80 taken as the standard of adequacy. A p-value of < 0.05 is taken as the criteria for the test result to be statistically significant and data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-85 years' old
* Both male and female patients
* ASA I-II
* Body mass index (BMI) ≤ 30 kg/m2
* Elective surgery under general anaesthesia with the use of laryngeal mask airway (LMA) / LMA Proseal / LMA Supreme
* Type of surgery: Urogynecological, General Surgery, Orthopedics, Eye, Vascular, Plastic
* Surgery/anaesthesia lasting for 0.5-3 hours

Exclusion Criteria:

* Patients with difficulty in swallowing, preexisting neuromuscular or central nervous system disorder
* Patients undergoing intra abdominal, thoracic, face, nasal or throat surgery
* Known condition interfering with gastric emptying
* Patients with cognitive or hearing impairment and inability to provide informed consent
* ASA III-IV patients
* Use of muscle relaxant during the course of general anesthesia
* Contraindication or previous adverse response to any of the study drugs

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The recovery of ability to swallow 20mls of water at designated time frame after response to command | up to 30 minutes after appropriate verbal response
  Patient is asked to swallow 20mls of water every 5 minutes after appropriate verbal response. Successful swallowing is defined as swallowing 20mls of water without drooling, coughing, choking or nausea. If patient fails to swallow at the first 5 minutes, the test will be repeated every 5 minutes until 30 minutes are up or until patient is able to swallow successfully

SECONDARY OUTCOMES:
Emergence and immediate recovery times after discontinuation of sevoflurane versus desflurane | A stopwatch will be used to record the time (in minutes) of patient obeying verbal command
  Emergence and immediate recovery times are the time taken by patient to open eyes to call or grip the observer's hands, and obey simple commands ie state his/her name or state his/her date of birth. A Stopwatch is used to record the time from discontinuation of the anaesthetic agent used to the emergence and immediate recovery times

CONTACTS AND LOCATIONS:
Overall Officials: Lee Fenky, MBBS (IMU), Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Mckay RE, Large MJC, Balea MC, Mckay WR. Airway reflexes return more rapidly after desflurane anesthesia than after sevoflurane anesthesia. Anesth Analg. 2005 Mar;100(3):697-700. doi: 10.1213/01.ANE.0000146514.65070.AE. PMID 15728054